CLINICAL TRIAL: NCT05658575
Title: A Multi-Center Phase 2/3 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Safety and Efficacy Study of Dapansutrile Tablets in Subjects With an Acute Gout Flare
Brief Title: Study of Dapansutrile Tablets in Subjects With an Acute Gout Flare
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLT1177-08
Record Dates: First submitted 2022-11-29; First posted 2022-12-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Gout Flare; Gout Attack; Gout Flare; Gouty Arthritis; Gout; Arthritis; Joint Pain
Keywords: gout; gouty arthritis; mono-articular arthritis; NLRP3; NLRP3 inhibitor; dapansutrile; OLT1177; joint pain; inflammation; gouty Inflammation; inflammasomes; IL-1 beta; IL-1 inflammation; autoinflammatory conditions; hyperuricemia; uric acid crystal; flare; small-molecule; therapeutic
MeSH Terms: conditions — Arthritis, Gouty; Gout; Arthritis; Arthralgia; Inflammation; Hyperuricemia | interventions — dapansutrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapansutrile (Experimental): An initial loading dose of 2000 mg dapansutrile on Day 1 followed by a maintenance regimen of 1000 mg dapansutrile twice daily starting 12 hours later through the second dose on Day 7, inclusive.
  Interventions: Drug: Dapansutrile
- Placebo Tablet (Placebo Comparator): An initial loading dose of matching placebo (to mimic dapansutrile dosing) on Day 1 followed by a maintenance regimen of matching placebo twice daily starting 12 hours later through the second dose on Day 7, inclusive.
  Interventions: Other: Placebo Tablet

INTERVENTIONS:
Drug: Dapansutrile — An initial loading dose of 2000 mg dapansutrile on Day 1 followed by a maintenance regimen of 1000 mg dapansutrile twice daily starting 12 hours later through the second dose on Day 7, inclusive.
  Other Names: OLT1177
  Arms: Dapansutrile
Other: Placebo Tablet — An initial loading dose of matching placebo (to mimic dapansutrile dosing) on Day 1 followed by a maintenance regimen of matching placebo twice daily starting 12 hours later through the second dose on Day 7, inclusive.
  Arms: Placebo Tablet

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of dapansutrile (OLT1177®) tablets in subjects with an acute gout flare.

DETAILED DESCRIPTION:
This is a multi-center Phase 2/3 randomized, double-blind, placebo-controlled, parallel-group safety and efficacy study of dapansutrile (OLT1177®), a specific NLRP3 inhibitor, conducted in subjects with acute gout flare. Up to 300 eligible subjects will be randomized 2:1 to one of two treatment arms to receive either dapansutrile tablets or matching placebo twice daily for 7 days. An initial loading dose on Study Day 1 will be followed by a twice daily maintenance dosing regimen.

Subjects presenting with acute gout flare that began within 96 hours prior to the Baseline/Day 1 visit will be evaluated for eligibility. Subjects who are determined to be eligible will be randomized into either an active treatment arm (2/3 of the subjects enrolled) or the placebo arm (1/3 of the subjects enrolled).

Eligible subjects who are randomized into the study will also be provided with rescue medication at the Baseline/Day 1 Visit. No other pain medications, anti-inflammatory drugs (e.g., steroids or nonsteroidal anti-inflammatory drugs), or treatments for gout flare are allowed during the Treatment Period.

During the Treatment Period, subjects will return to the clinic trial site on Day 4 and, following the 7-day Treatment Period, subjects will return to the clinical trial site on Day 8, and then Day 15 with safety data collected through Day 36.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 or older
* Clinical diagnosis of gout according to the 2015 ACR/EULAR Gout Classification Criteria:

A) Diagnosis of gout must be confirmed in the target joint as indicated by either the presence of monosodium urate (MSU) crystals by microscopic evaluation of synovial fluid from the target joint or bursa OR by imaging evidence of urate deposition in the target joint or bursa at the Screening/Baseline Visit/Study Day 1, or

B) Documented history in the target joint or bursa ; or documented history of 2 or more gout flares in the previous 18 months

* Confirmation of a gout flare in the target joint that began within 96 hours prior to the Screening/Baseline Visit
* Provide written informed consent and understand and comply with all trial requirements

Exclusion Criteria:

* Presence of any palpable and visible tophi by physical examination
* Has ≥ 4 joints with an acute gout flare at Screening/Baseline
* Presence of active rheumatoid arthritis or other acute inflammatory arthritis
* Evidence/suspicion of infectious/septic arthritis
* Clinically significant general pain or non-gout-related joint pain that would interfere with the subject's ability to accurately assess pain in the target joint
* Known diagnosis of chronic kidney disease or known history of renal impairment
* Positive test for severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) infection, if tested, within 4 weeks of the Screening/Baseline
* Active malignancy or recent malignancy with any systemic anti-cancer treatment
* Has a hypersensitivity or allergy to OLT1177® or other drugs in its class
* Hypersensitivity or allergy to paracetamol/acetaminophen
* Use of any prohibited concomitant medications/therapies over the periods defined in the protocol or planned use of any prohibited concomitant medications/therapies during the Treatment Period (including the use of paracetamol/acetaminophen within 4 hours prior to the Screening/Baseline Visit or other pain medications within 12 hours prior to the Screening/ Baseline Visit
* Use of any product containing paracetamol/acetaminophen within 4 hours prior to the Screening/Baseline Visit or planned use during the Treatment Period (with the exception of study-provided Rescue Medication [paracetamol/acetaminophen], which is permitted after completion of the first target joint pain assessment on Study Day 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of dapansutrile as an acute gout flare treatment compared to placebo in reducing joint pain at 72 hours post initial loading dose of IMP | 72 hours
  Change from baseline in the subject-assessed pain intensity score evaluated on a 100-mm visual analogue scale (VAS) in the target joint at 72 hours post initial loading dose for dapansutrile compared to placebo. The visual analog scale has anchors of 0 indicating no pain and 100 indicating the worst pain.

SECONDARY OUTCOMES:
Change in joint pain in the target joint at scheduled time points post initial loading dose of study drug | 12, 24, 36, 48 and 60 hours; 8 and 15 days
  Change from baseline in the subject-assessed pain intensity score evaluated on a 100-mm visual analogue scale (VAS) in the target joint at specified timepoints up to Day 15 post initial loading dose of study drug. The visual analog scale has anchors of 0 indicating no pain and 100 indicating the worst pain.
To assess the clinical activity of dapansutrile compared to placebo in treating signs and symptoms of an acute gout flare other than pain (tenderness, swelling, erythema, warmth, and range of motion). | 4 and 8 days
  Patient Global Assessment of Response to Treatment (PGART) will be completed by the subject through Day 8. The PGART is a 5-level Likert-type single item (i.e., one general question the Subject is asked to answer) about the overall perceived status of their response to treatment on a scale from "None" to "Excellent".
To assess the clinical activity of dapansutrile compared to placebo in treating signs and symptoms of an acute gout flare other than pain (tenderness, swelling, erythema, warmth, and range of motion) | 8 and 15 days
  Change from baseline in the Investigator-assessed Target Joint Score at scheduled assessments through Study Day 15. The Investigator-assessed Target Joint Score is a combined assessment of individual assessments for the following outcome domains: tenderness, swelling, erythema, warmth, and range of motion each with a scale of 0 through 3, with lower scoring in each domain indicating better outcomes in the respective domain.
To assess the clinical activity of dapansutrile compared to placebo in treating signs and symptoms of an acute gout flare other than pain (tenderness, swelling, erythema, warmth, and range of motion). | 4 and 8 days
  Investigator Global Assessment of Response to Treatment (IGART) will be completed by the Investigator through Study Day 8. The IGART is a 5-level Likert-type single item (i.e., one general question the Investigator is asked to answer) about the overall perceived status of the subject's response to treatment on a scale from "None" to "Excellent".
To further assess the clinical activity of dapansutrile compared to placebo in reducing joint pain at scheduled time points post initial loading dose of IMP. | 48 and 72 hours; 8 and 15 days
  Proportion of subjects with a response (defined as a 20%, 50%, or 70% reduction from baseline without using Rescue Medication) in the subject-assessed pain intensity score (100-mm VAS) in the target joint up to Day 15 post initial loading dose of study drug.
To assess the clinical activity of dapansutrile compared to placebo in treating signs and symptoms of an acute gout flare other than pain (tenderness, swelling, erythema, warmth, and range of motion). | 15 days
  Change from baseline in the subject-assessed Quality of Life (QoL) questionnaire Short Form Health Survey-12 version 2.0 (SF-12v2) at scheduled assessments through Study Day 15.
To further assess the clinical activity of dapansutrile compared to placebo in reducing joint pain at scheduled time points post initial loading dose of IMP. | 4, 8 and 15 days
  Change from baseline in the subject-assessed pain intensity score evaluated on a 100-mm visual analogue scale (VAS) in any actively flaring non-target joint(s) up to Day 15 post initial loading dose of study drug. The visual analog scale has anchors of 0 indicating no pain and 100 indicating the worst pain.
To characterize the population PK of dapansutrile and exposure-response relationship for efficacy and safety. | up to 15 days
  Blood samples will be drawn and analyzed in order to characterize the population PK of dapansutrile
Physical examinations | Up to 15 days
  Physical examinations will be conducted to assess changes in subject health throughout the duration of the study.
Vital signs | Up to 15 days
  Vital signs consisting of pulse, resting blood pressure, temperature and respirations will be recorded and analyzed for changes throughout the duration of the study
Electrocardiograms | 15 days
  Electrocardiograms will be captured and analyzed for changes throughout the duration of the study.
Safety laboratory measurements | Up to 15 days
  Blood samples will be drawn and analyzed for routine chemistry blood markers, routine hematology/complete blood count and routine urinalysis will be performed throughout the duration of the study
Adverse events | Up to 36 days
  Adverse events will be described with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the event.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates - Glendale, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates (AARA), P.C. - Mesa, Mesa, Arizona
  - American Institute of Research, Los Angeles, California
  - TriWest Research Associates, San Diego, California
  - Valiance Clinical Research - Tarzana, Tarzana, California
  - Hillcrest Medical Research, DeLand, Florida
  - SIMEDHealth, Gainesville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Arthritis Center of North Georgia - Gainesville, Gainesville, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Advanced Quality Medical Research, Orland Park, Illinois
  - The Research Group of Lexington, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Montana Medical Research, Missoula, Montana
  - NYU Langone, New York, New York
  - IMA Clinical Research - Manhattan, New York, New York
  - Altoona Research, Duncansville, Pennsylvania
  - Lower Country Rheumatology - Summerville, Summerville, South Carolina
  - Amarillo Center of Clinical Research, Amarillo, Texas
  - Utah Health - University of Utah Hospital, Salt Lake City, Utah
  - Clinical Trial Site, Bothell, Washington
  - Arthritis Northwest, Spokane, Washington
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital Saint Philibert, Lomme
  - Hôpital Lariboisière, Paris
  - CHU de Rouen - Hôpital Charles-Nicolle, Rouen
- Israel (4):
  - Emek Medical Center, Afula
  - Carmel Medical Center, Haifa
  - Rabin Medical Center - Beilinson and Hasharon, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Netherlands (3):
  - Reade Research BV, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
  - VieCuri Medisch Centrum, Venlo
- Spain (4):
  - Hospital Universitario san Juan de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid